CLINICAL TRIAL: NCT06702722
Title: Enhanced Problem-solving Therapy and HIV Engagement Support to Improve Perinatal Mental Health and HIV Outcomes in Malawi: A Randomized Controlled Trial
Brief Title: Enhanced Problem-solving Therapy and HIV Engagement Support to Improve Perinatal Mental Health & HIV Outcomes in Malawi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-0690; R01MH134660 (NIH)
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: HIV; Depression; Depression, Postpartum
MeSH Terms: conditions — Depression; Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: 2-arm individually randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Friendship Bench (Experimental): Friendship Bench problem-solving therapy, social support sessions and home visits during the 3rd trimester as well as postpartum.
  Interventions: Behavioral: Enhanced Friendship Bench
- Enhanced usual care (Active Comparator): Continue with usual outpatient care, enhanced to provide a mental health evaluation; brief supportive counseling; information, education, and support on common mental disorders; and (if indicated) facilitation of referral for further follow-up at a mental health clinic or psychiatric unit.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Enhanced Friendship Bench — Friendship Bench problem-solving therapy involving 4 prenatal and 2 postnatal counseling sessions, enhanced for HIV care engagement with 2 social support building sessions and monthly home visits for ART delivery and counseling during the 3rd trimester and the first 3 months postpartum.
  Arms: Enhanced Friendship Bench
Behavioral: Enhanced usual care — Usual care for mental health in public facilities in Malawi includes options for basic supportive counseling by a primary provider or nurse, medication management by the primary provider (amitriptyline is the one antidepressant typically available at primary health centers and is rarely prescribed for depression), referral to the clinic psychiatric nurse or mental health clinic, or in more severe cases referral to the psychiatric units at tertiary care hospitals. For the proposed study, usual care will be enhanced to provide a mental health evaluation; brief supportive counseling; information, education, and support on common mental disorders; and (if indicated) facilitation of referral for further follow-up at a mental health clinic or psychiatric unit.
  Arms: Enhanced usual care

SUMMARY:
The main objective of the proposed study is to evaluate the effectiveness of the Enhanced Friendship Bench intervention to improve perinatal depression, HIV care engagement, and infant health outcomes among pregnant women with HIV and depression in Malawi.

DETAILED DESCRIPTION:
In our R34 pilot trial, the Enhanced Friendship Bench intervention showed strong feasibility, acceptability, fidelity, and preliminary effectiveness to improve perinatal depression and engagement in HIV care. The goal of this proposal is to evaluate the effectiveness of the Enhanced Friendship Bench in a fully powered randomized control trial to improve perinatal depression, HIV care engagement, and infant health outcomes, examine mediators and moderators that help elucidate mechanisms of action, and collect key implementation measures to accelerate the translation of findings into practice.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for antenatal care at one of our 5 recruitment sites
* ≥ 18 years of age
* ≤ 34 weeks gestation
* HIV-positive, based on medical records
* Initiating, re-initiating, or on established ART during index pregnancy
* Elevated depressive symptoms as indicated by a EPDS score ≥10. The EPDS is widely used to assess perinatal mood disorders that has been validated in perinatal populations in Malawi with this cut point to identify probable perinatal depression

Exclusion Criteria:

* Suicidal ideation evaluated as acute risk.
* Other health concerns requiring emergent response.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive Symptoms | 6 months post partum
  Depressive symptoms at baseline and 6 months post partum will be evaluated via the Edinburgh Postnatal Depression Scale (EPDS). This screening instrument is a 10-item self-rating questionnaire with scores ranging from 0-30. Higher scores identify women who may be experiencing symptoms of perinatal depression. The scale is designed for use during pregnancy as well as the postpartum period, making it a versatile tool in maternal health care. Change in EPDS scores will be considered the primary outcome because this measure is specific to a perinatal population.
  The change in depressive symptoms from baseline to 6 months postpartum will be calculated as Baseline EPDS total score minus the 6 month post partum EPDS total score.
HIV Care Retention | 6 months post partum
  Retention in HIV care will be defined as ≥2 HIV visits that are at least 30 days apart in the first 6 months post-delivery; AND at least one visit in the first 90 days post-delivery and at least one visit in the second 90 days post-delivery. This definition is based on the minimum expected HIV care appointment schedule per Malawi HIV clinical guidelines. COVID-19 led to an enduring shift in ART prescribing patterns in Malawi, with many clinics moving from dispensing a 30-day ART supply to dispensing a 90-day supply in an effort to de-densify clinics. Consequently, two clinic visits in a 6-month period are typically sufficient to ensure continuous ART supply. While other retention measures such as the Missed or Kept Visit Proportion have high relevance in the US, they are less applicable in Malawian health care where missed visits are typically not recorded and only the dates of kept visits are noted in the medical record.

SECONDARY OUTCOMES:
Change in Depressive Symptoms | 6 months post partum
  Depressive symptoms will be measured at baseline and 6 months post partum using the Patient Health Questionnaire-9 (PHQ-9) which is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression with scores ranging from 0 to 27 where higher scores indicate greater self-reported depression. The change in depressive symptom scores from baseline to 6 months postpartum is calculated as baseline PHQ-9 score minus the 6 month post partum PHQ-9 score.
Proportion of patients achieving depression remission | 6 months post partum
  Depression remission will be defined as the proportion of patients who achieve depression remission at 6 months post partum.
  Depressive symptoms will be measured at 6 months post partum using the Patient Health Questionnaire-9 (PHQ-9) which is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression with scores ranging from 0 to 27 where higher scores indicate greater self-reported depression. Depression remission is defined as achievement of no or minimal depressive symptoms as defined by the widely used definition of a PHQ-9 score <5 at 6 months follow-up.
Proportion of patients achieving HIV viral suppression | 12 months post partum
  A secondary outcome for maternal HIV care engagement will be the proportion of patients with viral load suppression at 12 months. Viral load suppression will be defined as HIV RNA level <1000 copies/mL, the standard definition in Malawian medical care based on dried blood spot thresholds.
Infant Growth: height-for-age | 6 months post partum
  A secondary outcome for infant health will be infant growth at 6 months, defined as WHO z-score of height-for-age. This refers to a standardized score calculated using a child's measured height, weight, and age compared to the reference population established by the World Health Organization (WHO).
Infant Growth: weight-for-age | 6 months post partum
  A secondary outcome for infant health will be infant growth at 6 months, defined as WHO z-score of weight-for-age. This refers to a standardized score calculated using a child's measured height, weight, and age compared to the reference population established by the World Health Organization (WHO).
Infant Growth: weight-for-height | 6 months post partum
  A secondary outcome for infant health will be infant growth at 6 months, defined as WHO z-score of weight-for-height. This refers to a standardized score calculated using a child's measured height, weight, and age compared to the reference population established by the World Health Organization (WHO).

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pence, PhD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (5):
- Malawi (5):
  - Area 18 Health Center, Lilongwe
  - Area 25 Health Center, Lilongwe
  - Bwaila Hospital, Lilongwe
  - Kawale Health Center, Lilongwe
  - Likuni Mission Hosptial, Lilongwe

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill (UNC).
  Deidentified data will also be posted to the NIMH Data Archive pursuant to the requirements of that site.
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.